CLINICAL TRIAL: NCT02098096
Title: Development of a Negative Work Exercise Regimen as an Intervention for Posttraumatic Osteoarthritis of the Knee
Brief Title: Negative Work Exercise for the Treatment of Knee Arthritis
Acronym: PTOA-ECC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Harris-Love, Primary Investigator, Washington D.C. Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRB01625
Record Dates: First submitted 2014-03-19; First posted 2014-03-27 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis; Arthritis
Keywords: knee; arthritis; Veterans; strength; exercise; muscle
MeSH Terms: conditions — Osteoarthritis; Arthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Negative Work (Experimental): Negative work exercise via isokinetic knee extension/flexion will be performed twice per week for 12 weeks.
  Interventions: Other: Negative Work
- Stretching (Placebo Comparator): A home exercise program consisting of stretches for the major lower extremity muscles groups will be performed twice per week for 12 weeks.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Negative Work — Exercise will be performed twice per week for 12 weeks and exercise intensity will be progressed in three phases. These phases are:
  1. Familiarization
  2. Acclimatization
  3. Progression
  Exercise volume will be 3 sets of 10 repetitions (progressing to 4 sets at Week 6) for the knee flexors and extensors.
  All exercise will be supervised by a physical therapist and performed on a Biodex isokinetic dynamometer.
  Other Names: Eccentric exercise
  Arms: Negative Work
Other: Stretching — Home exercise program will be performed by the Placebo Comparator group and feature stretching over the 12 week intervention period.
  Arms: Stretching

SUMMARY:
The purpose of this study is to develop a negative work exercise regimen as an intervention for posttraumatic osteoarthritis (PTOA). "Negative work" is the force produced by muscles as they lengthen, and regularly occurs with common activities such as lowering an object from a shelf or walking down stairs. In this study, the investigators are examining the effectiveness of negative work exercise over a 12-week period in older, male, Veterans.

DETAILED DESCRIPTION:
Purpose: To develop a negative work exercise regimen as an intervention for posttraumatic osteoarthritis (PTOA). Given that the medical management of chronic PTOA is similar to idiopathic OA, the investigators propose a randomized, clinical trial to pilot negative work exercise in Veterans with knee OA as a proof-of-concept study for a subsequent investigation for people with PTOA.

Research Setting: DC VAMC, Physical Medicine & Rehabilitation Laboratory

Participants: Men between the ages of 50 and 70 years with a history of bilateral knee osteoarthritis will be consecutively recruited from the DC VAMC Rheumatology Service, Geriatrics Service, and Primary Care Medical Service.

Implications/Significance: The use of negative work exercise to enhance the force attenuation properties of muscle is an innovative approach to the treatment of OA and PTOA, and represents a significant departure from previous rehabilitation studies concerning arthritis. Use of a negative work paradigm may prove to be beneficial for older Veterans with OA and active military personnel with PTOA since similar muscle mechanics are involved in the energy absorption at the knee joint during gait. Despite the functional importance of lengthening muscle actions in protecting weight-bearing joints affected by arthritis, the authors are not aware of a study that involves the sole use of a negative work intervention for OA or PTOA. Addressing the aims of this proposal would lay the ground work needed to justify larger clinical trials featuring the negative work paradigm for soldiers with PTOA.

ELIGIBILITY:
Inclusion Criteria:

* Adult men 50 y.o. 70 years old will be recruited for this proposed study.
* Participant inclusion criteria includes having bilateral knee OA (Kellgren-Lawrence Grade 2 or 3) and sedentary (e.g., have not engaged in 3 exercise sessions per week for 3 consecutive months).
* Gait aides and orthoses will not preclude participation in this study.

Exclusion Criteria:

* Exclusion criteria include uncontrolled cardiovascular disease, non-ambulatory status, neurogenic weakness, knee extensor and flexor manual muscle test < 3 out of 5, lower extremity amputation, and current participation in a supervised exercise program.
* In addition, major surgical procedures within the last six months, unstable joints, endocrine or metabolic disorders that result in excessive fatigue or muscle weakness, or use of medications that may impair exercise tolerance would also preclude participation in this study.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-03; Primary Completion 2017-10 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Voluntary Contraction (MVC; ft-lbs) | 12 weeks
  Isokinetic assessment of MVC for the knee extensors and flexors.
Muscle thickness (cm) | 12 weeks
  Diagnostic ultrasound assessment of the rectus femoris

SECONDARY OUTCOMES:
Step Up/Over Test (movement time (s); kinetics (force indices) | 12 weeks
  The Step Up/Over Test involves stepping over an 8'' block with the use of a force plate. We will assess concentric force upon ascent, and eccentric force upon descent; the symmetry of these forces will be expressed as an index.
Physical Performance Test (PPT-7) | 12 weeks
  The PPT-7 is a performance-based assessment of function validated for use in older adults. Participant scores will be compared to reference, age-matched, data.
Knee injury and Osteoarthritis Outcome Score (KOOS; English version LK1.0) | 12 weeks
  Knee OA-specific questionnaire concerning mobility and health-related quality of life changes over time. Participant scores will be compared to a normative comparison group, and the published minimal detectable change scores as validated for a knee OA reference group.
Visual Analog Scale for Pain (VAS; 0-10) | 12 weeks
  VAS will be assessed using a pressure algometer at the mid-thigh before and after negative work exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, DSc, Principal Investigator — Washington DC VA Medical Center
Locations (1):
- Washington DC VA Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Harris-Love MO. Safety and efficacy of submaximal eccentric strength training for a subject with polymyositis. Arthritis Rheum. 2005 Jun 15;53(3):471-4. doi: 10.1002/art.21185. No abstract available. PMID 15934111
- [Background] Hernandez HJ, McIntosh V, Leland A, Harris-Love MO. Progressive Resistance Exercise with Eccentric Loading for the Management of Knee Osteoarthritis. Front Med (Lausanne). 2015 Jul 9;2:45. doi: 10.3389/fmed.2015.00045. eCollection 2015. PMID 26217665